CLINICAL TRIAL: NCT01255046
Title: A Phase II Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of STA-1 as an Add-on Treatment to Donepezil in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study of STA-1 as an Add-on Treatment to Donepezil
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinphar Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCCD09009A
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil plus STA-1 (Active Comparator)
  Interventions: Drug: Donepezil,; Drug: STA-1
- Donepezil plus placebo (Placebo Comparator)
  Interventions: Drug: Donepezil,; Drug: placebo

INTERVENTIONS:
Drug: Donepezil, — 10mg/tab, 1 tab/day for 72 weeks
Drug: STA-1 — 300mg/tab, 2 tab/tid for 72 weeks
  Arms: Donepezil plus STA-1
Drug: placebo — 2 tab/tid for 72 weeks
  Arms: Donepezil plus placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of STA-1 vs placebo as an add-on treatment to donepezil in patients with mild to moderate Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 50 years;
* Probable Alzheimer's disease diagnosed by the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria;
* MMSE score between 10-26, inclusive;
* Patient has been treated with donepezil 10 mg per day for at least 3 months prior to screening;
* Patient able to participate in all study evaluations and ingest oral medication as indicated;
* Patient has a responsible caregiver who will accompany the patient to all clinic visits during the study;
* Patient and the responsible caregiver have provided written informed consent before undergoing any study procedures.

Exclusion Criteria:

* Brain image (computed tomography (CT) scan or Magnetic Resonance Imaging (MRI) done within past 12 months prior to the study) and laboratory tests to exclude secondary dementia or non-Alzheimer's dementia;
* Patient with significant clinically central nervous system illness other than AD (e.g. Parkinson's disease, Human Immunodeficiency Virus (HIV) induced dementia, Hachinski Ischaemic Score (HIS) >4) or dementia complicated by other organic disease or delirium;
* Patient with a severe or uncontrolled Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Axis I disorder other than Alzheimer's disease, including amnestic disorders, schizophrenia or schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic, or post-traumatic stress disorder;
* Patient suffering from cerebral disturbances following a stroke or a cerebral trauma (if the event occurred within the last 6 months);
* Patient with a history of hypersensitivity to study drugs;
* Patient who has a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine (e.g., Addison's Disease), immune, neurologic, or hematologic disease as determined by the clinical judgment of the investigator;
* Participation in any research study within the last 30 days;
* Patient with significant alcohol or drug abuse as judged by the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ADAS-cog at Week 72 | from baselline (Visit 2) to week 72 (Visit 9)

SECONDARY OUTCOMES:
Change from baseline in Mini-Mental State Examination Scale Score (MMSE) at 72 week | baseline (V2) to week 72 (Visit 8)

CONTACTS AND LOCATIONS:
Overall Officials: Giia-Sheun Peng, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan